CLINICAL TRIAL: NCT06681597
Title: The Effect of Raspberry Ketone Intake on Plasma FGF21 Levels
Brief Title: Raspberry Ketone Intake Upregulates Circulating FGF21 and Induces Energy Expenditure in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanchang University (Other)
Responsible Party: Principal Investigator, Ting Luo, Professor, Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: I-MRER [2023] No. 68
Record Dates: First submitted 2024-11-02; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Diabetes; NAFLD (Nonalcoholic Fatty Liver Disease)
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — raspberry ketone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Human administrated with raspberry ketone (Experimental)
  Interventions: Dietary Supplement: Raspberry ketone
- Human administrated with placebo (Experimental)
  Interventions: Dietary Supplement: Raspberry ketone

INTERVENTIONS:
Dietary Supplement: Raspberry ketone — Human consumed 500mg of raspberry ketone

SUMMARY:
To investigate the molecular mechanism of raspberry ketone on regulating obesity, the investigators studied the effect of raspberry ketone intake on FGF21 in plasma.

The age of the volunteers were 18-60 years old, both male and female, without diabetes, hypertension and other diseases.

After ingestion of raspberry ketone (500mg), 2ml of blood was collected at 0 hours, 3 hours and 6 hours , and the FGF21 content in plasma was measured using a commercial reagent kit.

In addition, the investigators also studied the effect of raspberry ketone intake on energy metabolism 0 hours, 0.5 hours, 3 hours and 6 hours after consuming raspberry ketone (500mg).

ELIGIBILITY:
Inclusion Criteria:

No drugs were taken before the human study

Exclusion Criteria:

Patients with hypertension

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Impact of raspberry ketone consumption on plasma FGF21 level | Through study completion, an average of 1 year
Impact of raspberry ketone consumption on energy expenditure | Through study completion, an average of 1 year
  The oxygen consumption, heart rate, carbon dioxide production were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Background] Lopez HL, Ziegenfuss TN, Hofheins JE, Habowski SM, Arent SM, Weir JP, Ferrando AA. Eight weeks of supplementation with a multi-ingredient weight loss product enhances body composition, reduces hip and waist girth, and increases energy levels in overweight men and women. J Int Soc Sports Nutr. 2013 Apr 19;10(1):22. doi: 10.1186/1550-2783-10-22. PMID 23601452